CLINICAL TRIAL: NCT04729894
Title: Evaluating the Impact of a Safe Medication Storage Device on Modifiable Storage Behaviors and Pediatric Poisonings
Brief Title: Evaluating the Impact of a Safe Medication Storage Device
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Binghamton University (Other)
Collaborators: State University of New York - Upstate Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00002619
Record Dates: First submitted 2020-10-14; First posted 2021-01-29 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Poisoning; Safety Issues; Accidents Injury
Keywords: pediatric poisonings; medication storage; safe medication storage
MeSH Terms: conditions — Poisoning; Accidental Injuries | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Safe Medication Storage Device + Education (Experimental)
  Interventions: Other: Medication Lockbox; Behavioral: Education
- Education (Active Comparator)
  Interventions: Behavioral: Education

INTERVENTIONS:
Other: Medication Lockbox — Participants will receive a medication lockbox to store medications in their home.
  Arms: Safe Medication Storage Device + Education
Behavioral: Education — Participants will receive information on safe medication storage practices.

SUMMARY:
Despite the initial success of the 1970s Poison Prevention Packaging Act, the incidence of pediatric medication poisonings in the United States remains high. Unintentional pediatric medication ingestions result in significant morbidity and are associated with substantial healthcare use and costs. A majority of these medication poisonings involve a caregivers' medication and are caused by modifiable unsafe storage behaviors. A better understanding of factors associated with pediatric poisonings and safe medication storage behaviors is needed to inform public health policy and develop targeted educational interventions. Furthermore, low-cost, scalable interventions that improve medication storage behaviors and reduce pediatric poisonings are necessary to address this ongoing preventable public health crisis.

In preliminary experiments, a baseline evaluation of caregivers demonstrated that they are unlikely to have a locked medication storage device in their home, but would be willing to use a locked device if one was available. Additionally, a follow-up assessment indicated that a majority of caregivers had used their medication over a one-month period. The latter feasibility assessment supports both caregiver willingness to use a safe storage device and demonstrates that a storage device can improve medication storage behaviors in the short-term.

Given these findings, we hypothesize that pediatric medication poisonings are due to improper storage, that medication storage behaviors are influenced by demographic and household specific factors, and that medication lockboxes improve safe medication storage behaviors and reduce pediatric poisonings. These hypotheses will be evaluated using the studies in the following Specific Aims: (1) to identify factors associated with pediatric poisonings, (2) to identify factors associated with medication storage behaviors, (3) to evaluate the effect of lockboxes on storage behaviors and pediatric poisonings.

Should this exploratory study reveal factors associated with increased risk for pediatric poisoning or with safe medication storage, and should safe medication storage interventions improve modifiable storage behaviors or show a reduction in pediatric poisonings, the results will be used to inform targeted public health campaigns and to develop a low-cost, scalable national program for improving safe medication storage and reducing pediatric poisonings.

ELIGIBILITY:
Inclusion Criteria:

* Primary caregivers of pediatric patients less than 6 years of age presenting to the emergency department
* Adults (at least 18 years of age) who are responsible for supervising at least one child under the age of 6 years in their residence
* Supervision of at least one child under the age of 6 years for at least 3.5 days per week on average

Exclusion Criteria:

* pediatric patients who are critically ill or unstable
* pediatric patients presenting due to a poisoning related incident
* caregivers who are unable or unwilling to provide consent
* caregivers who are non-English speaking.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Medication Storage Behaviors | 1 year
  Participants will be evaluated at regular intervals over a one year period to evaluate the impact of a medication box + education, compared to education alone, on their short and long-term medication storage behaviors. These storage behaviors include storage location in the home, storage device(s), storage location height, co-storage with non-medication items, and alternative storage locations.

SECONDARY OUTCOMES:
Pediatric Poisonings | 1 year
  The rate of pediatric poisonings will be evaluated within each group and compared.
Medication Adherence | 1 year
  Household medication adherence will be evaluated within each group and compared. Adherence will be measured using the validated eight-item Morisky Medication Adherence Scale (MMAS-8).

IPD SHARING:
Plan to Share IPD: Undecided